CLINICAL TRIAL: NCT02898077
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase 3 Study of Weekly Paclitaxel With or Without Ramucirumab (IMC-1121B) in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma, Refractory to or Progressive After First-Line Therapy With Platinum and Fluoropyrimidine
Brief Title: A Study of Paclitaxel With or Without Ramucirumab (LY3009806) in Participants With Gastric or Gastroesophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15244; I4T-CR-JVCR (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma
Keywords: Second line; Angiogenesis; Vascular endothelial growth factor receptor 2
MeSH Terms: interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 8 milligram/kilogram (mg/kg) Ramucirumab + 80 mg/square meter (mg/m²) Paclitaxel (Experimental): 8 mg/kg ramucirumab was administered as an intravenous infusion (IV) on days 1 and 15, in combination with 80 mg/m² paclitaxel administered by IV on days 1, 8, and 15 of every 28-day cycle.
  Participants may continue on treatment until discontinuation criteria were met.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel
- Placebo + 80 mg/m² Paclitaxel (Experimental): Placebo was administered at a volume equivalent to a dose of 8 mg/kg by IV on Days 1 and 15, in combination with 80 mg/m² paclitaxel administered by IV on Days 1, 8, and 15 of a 28-day cycle.
  Participants may continue on treatment until discontinuation criteria were met.
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: 8 milligram/kilogram (mg/kg) Ramucirumab + 80 mg/square meter (mg/m²) Paclitaxel
Drug: Paclitaxel — Administered IV
Drug: Placebo — Administered IV
  Arms: Placebo + 80 mg/m² Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy of the study drug known as ramucirumab in participants with gastric and gastroesophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group Performance Status (ECOGPS) of 0 or 1 at study entry.
* Have a histopathologically or cytologically confirmed diagnosis of gastric or gastroesophageal junction (GEJ) adenocarcinoma.
* Have metastatic disease or locally advanced, unresectable disease.
* Have at least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
* Have experienced documented objective radiographic or symptomatic disease progression during first-line therapy, or within 4 months after the last dose of first-line therapy with any platinum/fluoropyrimidine doublet for unresectable or metastatic disease.
* Have adequate organ function.
* Have urinary protein ≤1+ on dipstick or routine urinalysis.

Exclusion Criteria:

* Have undergone major surgery within 28 days prior to randomization.
* Have received any first-line chemotherapy other than platinum and fluoropyrimidine with or without anthracycline for advanced gastric or GEJ adenocarcinoma.
* Have received any previous systemic therapy (including investigational agents) targeting vascular endothelial growth factor (VEGF) or the VEGF receptor signaling pathways.
* Have a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to randomization.
* Have significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal (GI) tract within 3 months prior to study entry.
* Have a history of GI perforation and/or fistulae within 6 months prior to randomization.
* Have experienced any arterial thromboembolic event within 6 months prior to randomization.
* Have uncontrolled arterial hypertension (systolic blood pressure ≥160 millimeters of mercury [mmHg] or diastolic blood pressure ≥100 mmHg) despite standard medical management.
* Have a serious or nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to randomization.
* Have a serious illness or medical condition(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- China (20):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - First hospital affiliated to Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union (Xiehe) Hospital, Wuhan, Hubei
  - Wu Han Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nan Jing No. 81 Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hosp Affiliated Hosp of Nanjing Univ Med, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tang Du Hospital, The Second Teaching Hospital of FMMU, Xi’an, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- Malaysia (5):
  - Hospital Umum Sarawak, Kuching, Sarawak
  - Advanced Medical & Dental Institute HUSM, Kepala Batas, Pulau Pinang
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - National Cancer Institute, Wilayah Persekutuan
- Philippines (3):
  - Cebu Doctors Hospital, Cebu City, Cebu
  - Dr. Pablo O. Torre Memorial Hospital, Bacolod
  - De La Salle Health Sciences Institute, Cavite City
- Thailand (4):
  - Rajavithi Hospital, Bangkok, Ratchathewi District
  - King Chulalongkorn Memoiral Hospsital, Bangkok
  - Police General Hospital, Bangkok
  - Khon Kaen Hospital, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Xu RH, Zhang Y, Pan H, Feng J, Zhang T, Liu T, Qin Y, Qin S, Yin X, Liu B, Ba Y, Yang N, Voon PJ, Tanasanvimon S, Zhou C, Zhang WL, Shen L. Efficacy and safety of weekly paclitaxel with or without ramucirumab as second-line therapy for the treatment of advanced gastric or gastroesophageal junction adenocarcinoma (RAINBOW-Asia): a randomised, multicentre, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2021 Dec;6(12):1015-1024. doi: 10.1016/S2468-1253(21)00313-7. Epub 2021 Oct 7. PMID 34626550

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Participant Flow, participants who completed were those who died on treatment or during follow-up.
Period: Overall Study
Arm/Group | 8 Milligram/Kilogram (mg/kg) Ramucirumab + 80 mg/Square Meter (mg/m²) Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Started | 294 | 146
Received at Least 1 Dose of Study Drug | 293 | 145
Completed | 246 | 123
Not Completed | 48 | 23
Not completed — Enrolled/randomized, but never treated | 1 | 1
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Sponsor Decision | 32 | 13
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Discontinued from treatment but refused follow-up | 2 | 1
Not completed — Ended extension period | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel: 8 mg/kg ramucirumab was administered as an IV on days 1 and 15, in combination with 80 mg/m² paclitaxel administered by IV on days 1, 8, and 15 of every 28-day cycle.
  Participants may continue on treatment until discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel | Total
Number analyzed (Participants) | 294 | 146 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.00 (11.49) | 56.20 (11.12) | 56.10 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 50 | 139
  Male | 205 | 96 | 301
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 290 | 145 | 435
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 257 | 135 | 392
  Malaysia | 18 | 7 | 25
  Philippines | 6 | 2 | 8
  Thailand | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Time Frame: Randomization to the Date of the First Radiographically Documented Progressive Disease or Death from Any Cause (Up To 30 Months)
Population: All randomized participants. Censored participants: Ramucirumab +Paclitaxel = 67, Placebo + Paclitaxel = 16.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 294 | 146
Months | 4.14 [3.71 to 4.30] | 3.15 [2.83 to 4.14]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs Placebo + 80 mg/m² Paclitaxel; Test type: Superiority; p = 0.0184, Log Rank; Hazard Ratio (HR) = 0.765, 95% CI 2-sided [0.613 to 0.955]

2. Primary Outcome: Overall Survival (OS)
Description: OS defined as the time from randomization to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: Randomization to Date of Death from Any Cause (Up To 37 Months)
Population: All randomized participants. Censored participants: Ramucirumab +Paclitaxel = 52, Placebo + Paclitaxel = 25.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 294 | 146
Months | 8.71 [7.98 to 9.49] | 7.92 [6.31 to 9.10]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs Placebo + 80 mg/m² Paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.963, 95% CI 2-sided [0.771 to 1.203]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was time from the date of randomization to the date of radiographic progression (according to RECIST v.1.1). If a participant died due to any reason without radiographic progression, TTP is censored at the last adequate tumor assessment. Target lesions: Progressive Disease (PD): At least a 20% increase in the sum of diameters of lesions vs the smallest sum on study (the sum must also demonstrate an absolute increase of at least 5 mm); or the appearance of new lesion(s). Non target lesions: PD: Unequivocal progression of existing lesions or the appearance of new lesion(s).
Time Frame: Randomization to the Date of the First Radiographically Documented Progressive Disease (Up To 30 Months)
Population: All randomized participants. Censored participants: Ramucirumab +Paclitaxel = 98, Placebo + Paclitaxel = 36.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 294 | 146
Months | 4.27 [4.14 to 5.52] | 4.07 [2.92 to 4.17]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs Placebo + 80 mg/m² Paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.761, 95% CI 2-sided [0.598 to 0.968]

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Randomization to Objective Disease Progression (Up To 30 Months)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 294 | 146
Percentage of participants | 26.5 [21.6 to 32.0] | 21.9 [15.5 to 29.5]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs Placebo + 80 mg/m² Paclitaxel; Test type: Superiority; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.2]

5. Secondary Outcome: Duration of Objective Response (DoR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Date of Objective Response to the Date of the First Radiographically Documented Progressive Disease or Death Due to Any Cause (Up To 24 Months)
Population: All randomized participants with response. Censored participants: Ramucirumab +Paclitaxel = 1, Placebo + Paclitaxel = 4.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 78 | 32
Months | 4.34 [3.12 to 5.22] | 2.83 [2.56 to 4.14]
Statistical Analysis 1: Comparison: 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel vs Placebo + 80 mg/m² Paclitaxel; Test type: Superiority; Hazard Ratio (HR) = 0.905, 95% CI 2-sided [0.577 to 1.421]

6. Secondary Outcome: Best Change From Baseline on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures global health status, 5 functional domains (physical, role, cognitive, emotional, and social) and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, scores range from 0 to 100 with higher scores representing a better level of functioning. For symptoms scales, scores range from 0 to 100 with higher scores representing a greater degree of symptoms. Least square (LS) mean value of changing from baseline to short-term follow up was estimated from the mixed model that was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 20 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EORTC QLQ-C30 data at short term follow up for each EORTC QLQ-C30 items.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 272 | 133
Units on a scale
  Global health status | 5.30 (1.18) | 8.43 (1.56)
  Functional scale: Physical functioning | 1.09 (0.82) | 1.20 (1.10)
  Functional scale: Role functioning | 0.60 (1.13) | 1.27 (1.49)
  Functional scale: Emotional functioning | 5.89 (0.90) | 4.72 (1.19)
  Functional scale: Cognitive functioning | 2.87 (0.84) | 2.12 (1.11)
  Functional scale: Social functioning | 2.71 (1.19) | 2.98 (1.59)
  Symptom scale: Fatigue | -4.20 (1.14) | -5.63 (1.51)
  Symptom scale: Nausea and vomiting | -4.84 (0.77) | -3.80 (1.03)
  Symptom scale: Pain | -6.89 (1.07) | -7.01 (1.43)
  Symptom scale: Dyspnea | -2.18 (0.95) | -2.65 (1.27)
  Symptom scale: Insomnia | -5.73 (1.18) | -7.06 (1.57)
  Symptom scale: Appetite loss | -7.84 (1.30) | -10.26 (1.73)
  Symptom scale: Constipation | -6.35 (1.11) | -5.41 (1.48)
  Symptom scale: Diarrhea | -2.51 (0.86) | -3.03 (1.14)
  Symptom scale: Financial difficulties | -8.49 (1.60) | -8.12 (2.13)

7. Secondary Outcome: Worst Change From Baseline on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures global health status, 5 functional domains (physical, role, cognitive, emotional, and social) and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, scores range from 0 to 100 with higher scores representing a better level of functioning. For symptoms scales, scores range from 0 to 100 with higher scores representing a greater degree of symptoms. LS Mean value of changing from baseline to short-term follow up was estimated from the mixed model that was controlled for Treatment, visit, Treatment*Visit and baseline.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 20 Months)
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 272 | 133
Units on a scale
  Global health status | -14.42 (1.32) | -9.83 (1.75)
  Functional scale: Physical functioning | -14.31 (1.30) | -11.71 (1.73)
  Functional scale: Role functioning | -18.46 (1.72) | -14.39 (2.28)
  Functional scale: Emotional functioning | -9.80 (1.30) | -6.77 (1.72)
  Functional scale: Cognitive functioning | -13.66 (1.40) | -12.08 (1.85)
  Functional scale: Social functioning | -17.05 (1.73) | -16.52 (2.30)
  Symptom scale: Fatigue | 15.28 (1.36) | 10.17 (1.80)
  Symptom scale: Nausea and vomiting | 8.57 (1.46) | 8.66 (1.95)
  Symptom scale: Pain | 14.01 (1.50) | 10.11 (2.00)
  Symptom scale: Dyspnea | 16.58 (1.51) | 8.34 (2.01)
  Symptom scale: Insomnia | 14.14 (1.74) | 7.97 (2.32)
  Symptom scale: Appetite loss | 17.06 (1.85) | 11.11 (2.46)
  Symptom scale: Constipation | 8.39 (1.57) | 6.58 (2.08)
  Symptom scale: Diarrhea | 13.41 (1.39) | 5.67 (1.85)
  Symptom scale: Financial difficulties | 10.11 (1.80) | 9.32 (2.39)

8. Secondary Outcome: Change From Baseline in Participant-Reported European-Quality of Life-5 Dimension Instrument-3 Levels (EQ-5D-3L) Index Score
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. A regression equation defines a utility value for these health states to generate an index score. The possible values for index score range from -0.594 (severe problems in all 5 dimensions) to 1 (no problem in all dimensions) on a scale where 1 represents the best possible health state.
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 20 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 3L data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123 | 56
Units on a scale | -0.1351 (0.2472) | -0.1303 (0.1765)

9. Secondary Outcome: Change From Baseline in Participant-Reported EQ-5D-3L Visual Analog Scale (VAS) Score
Description: EQ-5D-3L is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each of which has 3 levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. The EQ-5D VAS is used to record a participant's rating for his/her current health-related quality of life state on the day of questionnaire administration and is captured on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, 30 Days After Treatment Discontinuation (Up To 20 Months)
Population: All randomized participants who received at least one dose of study drug with baseline and post-baseline EQ-5D 3L data.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
Number analyzed (Participants) | 123 | 56
millimeter (mm) | -9.6 (20.11) | -8.6 (15.88)

ADVERSE EVENTS:
Time Frame: Adverse Events: Randomization Up To 26 Months; All-Cause Mortality: Randomization to Date of Death from Any Cause (Up To 37 Months)
Description: Adverse events: All randomized participants who received at least 1 dose of study drug. Mortality: All randomized participants.
Arm/Group | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel | Placebo + 80 mg/m² Paclitaxel
All-Cause Mortality (participants affected / at risk) | 246/294 | 123/146
Serious Adverse Events (participants affected / at risk) | 100/293 | 37/145
Other Adverse Events (participants affected / at risk) | 287/293 | 143/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=293) | Placebo + 80 mg/m² Paclitaxel (N=145)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow toxicity (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (14) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (5) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (3)
Intestinal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 2 (2)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 5 (5)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (26) | 3 (3)
Platelet count decreased (Investigations) | 9 (10) | 0 (0)
White blood cell count decreased (Investigations) | 12 (21) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab + 80 mg/m² Paclitaxel (N=293) | Placebo + 80 mg/m² Paclitaxel (N=145)
Anaemia (Blood and lymphatic system disorders) | 195 (338) | 94 (161)
Leukopenia (Blood and lymphatic system disorders) | 17 (64) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 16 (59) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 47 (54) | 15 (17)
Abdominal pain (Gastrointestinal disorders) | 38 (45) | 26 (32)
Abdominal pain upper (Gastrointestinal disorders) | 27 (38) | 4 (4)
Ascites (Gastrointestinal disorders) | 16 (17) | 7 (7)
Constipation (Gastrointestinal disorders) | 50 (64) | 26 (30)
Diarrhoea (Gastrointestinal disorders) | 71 (111) | 21 (40)
Gingival bleeding (Gastrointestinal disorders) | 16 (24) | 1 (1)
Nausea (Gastrointestinal disorders) | 54 (67) | 22 (29)
Vomiting (Gastrointestinal disorders) | 51 (79) | 22 (27)
Fatigue (General disorders) | 28 (31) | 8 (9)
Influenza like illness (General disorders) | 9 (9) | 11 (14)
Malaise (General disorders) | 74 (94) | 37 (47)
Oedema peripheral (General disorders) | 35 (40) | 10 (10)
Pain (General disorders) | 20 (22) | 12 (18)
Pyrexia (General disorders) | 53 (72) | 24 (32)
Pneumonia (Infections and infestations) | 12 (14) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 25 (29) | 7 (7)
Urinary tract infection (Infections and infestations) | 9 (13) | 11 (14)
Alanine aminotransferase increased (Investigations) | 88 (160) | 31 (43)
Aspartate aminotransferase increased (Investigations) | 100 (216) | 35 (55)
Bilirubin conjugated increased (Investigations) | 7 (9) | 9 (12)
Blood alkaline phosphatase increased (Investigations) | 34 (53) | 17 (23)
Blood bilirubin increased (Investigations) | 65 (135) | 35 (57)
Blood creatinine increased (Investigations) | 13 (14) | 8 (10)
Blood lactate dehydrogenase increased (Investigations) | 9 (13) | 9 (14)
Gamma-glutamyltransferase increased (Investigations) | 36 (45) | 14 (21)
Lymphocyte count decreased (Investigations) | 27 (59) | 8 (13)
Neutrophil count decreased (Investigations) | 223 (892) | 102 (286)
Platelet count decreased (Investigations) | 88 (232) | 17 (29)
Weight decreased (Investigations) | 59 (75) | 22 (27)
White blood cell count decreased (Investigations) | 227 (926) | 107 (351)
White blood cell count increased (Investigations) | 6 (6) | 9 (12)
Decreased appetite (Metabolism and nutrition disorders) | 81 (99) | 32 (37)
Hyperglycaemia (Metabolism and nutrition disorders) | 27 (41) | 21 (38)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (21) | 8 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 90 (125) | 31 (53)
Hypocalcaemia (Metabolism and nutrition disorders) | 46 (64) | 14 (20)
Hypochloraemia (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 32 (44) | 15 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 31 (41) | 23 (28)
Hypophosphataemia (Metabolism and nutrition disorders) | 20 (46) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (41) | 14 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 8 (8)
Dizziness (Nervous system disorders) | 13 (16) | 8 (12)
Headache (Nervous system disorders) | 18 (25) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 36 (42) | 22 (25)
Paraesthesia (Nervous system disorders) | 26 (27) | 10 (11)
Insomnia (Psychiatric disorders) | 37 (47) | 11 (12)
Proteinuria (Renal and urinary disorders) | 99 (164) | 31 (57)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 9 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 (71) | 9 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 83 (88) | 55 (57)
Rash (Skin and subcutaneous tissue disorders) | 17 (21) | 3 (3)
Hypertension (Vascular disorders) | 66 (137) | 25 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02898077/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT02898077/SAP_001.pdf